CLINICAL TRIAL: NCT04021589
Title: A Study of Chemotherapy With WeiLeShu Versus Chemotherapy Alone in Patients With Metastatic Colorectal Cancer
Brief Title: Chemotherapy w/wo WeiLeShu in Metastatic Colorectal Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Zhejiang University (Other)
Responsible Party: Principal Investigator, Weijia Fang, MD, director, Zhejiang University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Microbio-WLS001
Record Dates: First submitted 2019-07-11; First posted 2019-07-16 (Actual); Last update posted 2023-01-30 (Actual); Status verified 2023-01

CONDITIONS: Microbial Colonization; Colorectal Cancer
MeSH Terms: conditions — Communicable Diseases; Colorectal Neoplasms | interventions — Drug Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- WLS-intervention group (Experimental): chemotherapy + WLS
  Interventions: Drug: Weileshu; Drug: Chemotherapy
- the control group (Active Comparator): chemotherapy
  Interventions: Drug: Chemotherapy

INTERVENTIONS:
Drug: Weileshu — a probiotics products which help to rebuild homeostasis of gut microbiome
  Arms: WLS-intervention group
Drug: Chemotherapy — chemotherapy

SUMMARY:
A total of 50 patients with metastatic colorectal cancer will be enrolled in the study. The patients were randomly divided into the WLS-intervention group and the control group. The two groups of patients were given the most appropriate medication according to the specific conditions of the disease. Patients in the intervention group received additional oral administration of Weileshu, a probiotics product (Tongchuang Biotechnology).

ELIGIBILITY:
Inclusion Criteria:

* At least 18 years of age, of any race or sex who are eligible to sign written consent and have undergone prior resection of histological evidence of colorectal cancer
* Hematologic function: ANC ≥ 1.5 x 10 /L, platelets ≥ 75 x 10 /L, and hemoglobin > 9 g/dL Adequate liver function as measured by: total bilirubin ≤ 2.0 mg/dl, AST and ALT ≤ 5 ULN, albumin ≥ 2.5 g/dl Adequate renal function as measured by: creatinine ≤ 2.9 mg/dl, > 50 ml/min calculated by the C-G equation Non-pregnant women of childbearing potential and fertile men are required to use effective contraception (negative pregnancy test for women of child-bearing age) ECOG status ≤ 1 at screening

Exclusion Criteria:

-

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2019-07-11 (Actual); Primary Completion 2021-10-30 (Actual); Study Completion 2021-10-30 (Actual)

PRIMARY OUTCOMES:
progression free survival | up to approximately half a year
  time from randomization to progression

SECONDARY OUTCOMES:
overall survival | up to approximately two years
  time from randomization to death

CONTACTS AND LOCATIONS:
Overall Officials: Weijia Fang, Doctor, Principal Investigator — First Affiliated Hospital of Zhejiang University
Locations (1):
- First affiliated hospital, Zhejiang University, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No